CLINICAL TRIAL: NCT02984774
Title: Does Telomerase Activity Have an Effect on Infertility in Patients With Endometriosis ? Assessment of Telomerase Activity in Eutopic, Ectopic Endometrial Tissue and Serum
Brief Title: Assessment of Telomerase Activity in Endometrial Tissue and Serum in Endometriosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nigar Sofiyeva, Resident Doctor, Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 53684
Record Dates: First submitted 2016-12-01; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Endometriosis Ovaries; Infertility, Female
Keywords: Endometriosis; Infertility; Telomerase activity
MeSH Terms: conditions — Infertility, Female; Endometriosis; Infertility | interventions — Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Infertile endometriosis (Experimental): Cystic wall segment from cystectomy material, endometrial sampling during the surgery and peripheric blood sampling during intravenous catheterization during anesthesia.
  Interventions: Procedure: Cystectomy; Procedure: Endometrial sampling; Procedure: Peripheric blood sampling
- Fertile endometriosis (Experimental): Cystic wall segment from cystectomy material, endometrial sampling during the surgery and peripheric blood sampling during intravenous catheterization during anesthesia.
  Interventions: Procedure: Cystectomy; Procedure: Endometrial sampling; Procedure: Peripheric blood sampling
- Control (Other): Ovarian tissue sampling, endometrial sampling from hysterectomy and oophorectomy pieces and peripheric blood sampling during intravenous catheterization during anesthesia.
  Interventions: Procedure: Endometrial sampling; Procedure: Peripheric blood sampling; Procedure: Ovarian tissue sampling

INTERVENTIONS:
Procedure: Cystectomy — Segment of cystic wall from the patients for planned cystectomy was taken after operation and was preserved at -80º Celsius for further analysis
  Arms: Fertile endometriosis; Infertile endometriosis
Procedure: Endometrial sampling — Endometrial sampling was performed at the same operation with the planned operation for the main indication and was preserved at -80º Celsius for further analysis
  Other Names: Pipelle endometrial suction curettage
Procedure: Peripheric blood sampling — 4 cc peripheric venous blood was sampled into the EDTA(Ethylenediaminetetraacetic acid)-containing tubes during catheterization for anesthesia was preserved at 4º Celsius for further analysis
Procedure: Ovarian tissue sampling — 2cm linear tissue sample from ovarian cortex was performed at the same operation with the planned operation for the main indication and was preserved at -80º Celsius for further analysis
  Arms: Control

SUMMARY:
The goal of the study was the detection of telomerase activity in eutopic, ectopic endometrial tissue and in peripheral blood and finding the correlation between the telomerase activity and clinic findings. With these results, confirmation of the hypothesis regarding the endometriosis pathogenesis and endometriosis-related infertility was aimed.

DETAILED DESCRIPTION:
Although distorted pelvic anatomy, impaired peritoneal, humoral and cellular functions, decreased implantation rate, oocyte and embryo quality, obstructed utero tubal connection are most researched aspects of endometriosis-related infertility, etiopathogenesis of endometriosis-related infertility still remains controversial.

Endometrial cell is a unique eukaryotic somatic cell with cyclic telomerase activity. Hormone-dependent cyclic variation of endometrial telomerase activity was stated in previous studies. On the other hand telomerase, activity was shown in endometriotic lesions, whereas this activity lacks in most of the somatic cells.

In this study, assessment of possible relation to increased telomerase activity in infertile patients with endometriosis was aimed.

Before published studies were assessed telomerase activity in benign and malign gynecological conditions and in endometriosis tissue, as well. But evaluation of ectopic and eutopic endometrial tissue and serum telomerase activity in infertile and fertile endometriosis and healthy control subjects was not performed.

Correlation of telomerase activity and endometriosis-related infertility was aimed in this study.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Infertility Clinical and histological diagnosis of endometriosis

Exclusion Criteria:

Malign disorders Hormone replacement treatment Oral Contraceptive using

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-06; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Telomerase activity | through study completion, an average of 1 year
  Assessment of telomerase activity with Telomeric Repeat Amplification Protocol Polymerase Chain Reaction method from tissue and blood

SECONDARY OUTCOMES:
Age in years | During admission to hospital for surgery
  From patient anamnesis
Marital status (single, married, divorced, widow) | During admission to hospital for surgery
  From patient anamnesis
Smoking status ( yes/no) | During admission to hospital for surgery
  From patient anamnesis
BMI in kg/m2 | During admission to hospital for surgery
  From patient anamnesis
Cystic size in cm | During operation
  Macroscopically assessment during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Engin Oral, MD, Study Director — Istanbul University
Locations (1):
- Nigar Sofiyeva, Istanbul, Non-US/Non-Canadian, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
General results is available for sharing.

REFERENCES:
- [Background] Schenken RS, Asch RH, Williams RF, Hodgen GD. Etiology of infertility in monkeys with endometriosis: luteinized unruptured follicles, luteal phase defects, pelvic adhesions, and spontaneous abortions. Fertil Steril. 1984 Jan;41(1):122-30. doi: 10.1016/s0015-0282(16)47552-7. PMID 6420199
- [Background] Bedaiwy MA, Falcone T, Sharma RK, Goldberg JM, Attaran M, Nelson DR, Agarwal A. Prediction of endometriosis with serum and peritoneal fluid markers: a prospective controlled trial. Hum Reprod. 2002 Feb;17(2):426-31. doi: 10.1093/humrep/17.2.426. PMID 11821289
- [Background] Pizzo A, Salmeri FM, Ardita FV, Sofo V, Tripepi M, Marsico S. Behaviour of cytokine levels in serum and peritoneal fluid of women with endometriosis. Gynecol Obstet Invest. 2002;54(2):82-7. doi: 10.1159/000067717. PMID 12566749
- [Background] Lebovic DI, Mueller MD, Taylor RN. Immunobiology of endometriosis. Fertil Steril. 2001 Jan;75(1):1-10. doi: 10.1016/s0015-0282(00)01630-7. PMID 11163805
- [Background] Genbacev OD, Prakobphol A, Foulk RA, Krtolica AR, Ilic D, Singer MS, Yang ZQ, Kiessling LL, Rosen SD, Fisher SJ. Trophoblast L-selectin-mediated adhesion at the maternal-fetal interface. Science. 2003 Jan 17;299(5605):405-8. doi: 10.1126/science.1079546. PMID 12532021
- [Background] Cunha-Filho JS, Gross JL, Bastos de Souza CA, Lemos NA, Giugliani C, Freitas F, Passos EP. Physiopathological aspects of corpus luteum defect in infertile patients with mild/minimal endometriosis. J Assist Reprod Genet. 2003 Mar;20(3):117-21. doi: 10.1023/a:1022625106489. PMID 12735387
- [Background] Kissler S, Hamscho N, Zangos S, Gatje R, Muller A, Rody A, Dobert N, Menzel C, Grunwald F, Siebzehnrubl E, Kaufmann M. Diminished pregnancy rates in endometriosis due to impaired uterotubal transport assessed by hysterosalpingoscintigraphy. BJOG. 2005 Oct;112(10):1391-6. doi: 10.1111/j.1471-0528.2005.00676.x. PMID 16167942
- [Background] Tanaka M, Kyo S, Takakura M, Kanaya T, Sagawa T, Yamashita K, Okada Y, Hiyama E, Inoue M. Expression of telomerase activity in human endometrium is localized to epithelial glandular cells and regulated in a menstrual phase-dependent manner correlated with cell proliferation. Am J Pathol. 1998 Dec;153(6):1985-91. doi: 10.1016/S0002-9440(10)65712-4. PMID 9846988
- [Background] Williams CD, Boggess JF, LaMarque LR, Meyer WR, Murray MJ, Fritz MA, Lessey BA. A prospective, randomized study of endometrial telomerase during the menstrual cycle. J Clin Endocrinol Metab. 2001 Aug;86(8):3912-7. doi: 10.1210/jcem.86.8.7729. PMID 11502832
- [Result] Kim CM, Oh YJ, Cho SH, Chung DJ, Hwang JY, Park KH, Cho DJ, Choi YM, Lee BS. Increased telomerase activity and human telomerase reverse transcriptase mRNA expression in the endometrium of patients with endometriosis. Hum Reprod. 2007 Mar;22(3):843-9. doi: 10.1093/humrep/del425. Epub 2006 Oct 31. PMID 17077107
- [Result] Hapangama DK, Turner MA, Drury JA, Quenby S, Saretzki G, Martin-Ruiz C, Von Zglinicki T. Endometriosis is associated with aberrant endometrial expression of telomerase and increased telomere length. Hum Reprod. 2008 Jul;23(7):1511-9. doi: 10.1093/humrep/den172. Epub 2008 May 2. PMID 18456668
- [Result] Lehner R, Enomoto T, McGregor JA, Shroyer AL, Haugen BR, Pugazhenthi U, Shroyer KR. Quantitative analysis of telomerase hTERT mRNA and telomerase activity in endometrioid adenocarcinoma and in normal endometrium. Gynecol Oncol. 2002 Jan;84(1):120-5. doi: 10.1006/gyno.2001.6474. PMID 11748987